CLINICAL TRIAL: NCT06141460
Title: A Phase I/IIa, Dose-escalation and Dose-extension Study to Evaluate the Safety and Efficacy of Single Subretinal Injection of RRG001 in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Safety and Efficacy of RRG001 Gene Therapy in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Refreshgene Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RRG001-101
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RRG001 Dose1 (Experimental): Frequency of administration: one time injection.
  Interventions: Drug: RRG001
- RRG001 Dose2 (Experimental): Frequency of administration: one time injection.
  Interventions: Drug: RRG001
- RRG001 Dose3 (Experimental): Frequency of administration: one time injection.
  Interventions: Drug: RRG001
- RRG001 Dose4 (Experimental): Frequency of administration: one time injection.
  Interventions: Drug: RRG001

INTERVENTIONS:
Drug: RRG001 — Administered via Subretinal injection. Dosage form: injection solution.

SUMMARY:
A Phase I/IIa, Dose-escalation and Dose-expansion Study to Evaluate the Safety and Efficacy of Single Subretinal Injection of RRG001 in Subjects With Neovascular Age-related Macular Degeneration

DETAILED DESCRIPTION:
This study adopts a multicenter, single-arm, open-label phase I/IIa seamless study design and comprises two stages, i.e., phase I 3+3 dose escalation study and a phase IIa dose expansion study. Four dose groups are preset for the phase I dose escalation study; 3-6 subjects will be enrolled for each dose group, and it is planned to enroll 12-24 subjects. The phase IIa dose expansion study will be conducted successively at the doses after safety assessments of dose 2 and/or dose 3 in phase I are completed. Twelve subjects are expected to be enrolled for each dose group, with a total of 24 subjects will be enrolled overall. The sponsor will assess whether or not to adjust the dose(s) and sample size for the exploration study based on the results in the phase I exploration study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are willing and able to follow study procedures.
* Patinets ≥50 years old.
* Clinically diagnosed with CNV secondary to nAMD.
* BCVA of the study eye is ≥5 letters and ≤73 letters(Snellen 20/800~20/40), as well as that of the other eye ≥19 letters(Snellen 20/400).
* Responding to anti-VEGF

Exclusion Criteria:

* Presence of any other eye diseases other than nAMD in study eye that would affect the treatment or confusing the interpretation of the study results , as judged by the investigator.
* CNV or macular edema in the study eye secondary to any causes other than AMD.
* Uncontrolled glaucoma.
* Uncontrolled hypertension despite medication.
* Pregnant or lactating women or individuals with reproductive potential who are unwilling to take effective contraception during the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Week 52
  incidence of AEs and SAEs

SECONDARY OUTCOMES:
Efficacy after RRG001 injection | Week 52
  change in best-corrected visual acuity (BCVA)；
Efficacy after RRG001 injection | Week 52
  change in central retinal thickness (CRT)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China